CLINICAL TRIAL: NCT00067860
Title: Diet/Growth Factor Mechanisms of Gut Adaptation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thomas R. Ziegler, MD, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00035030; R01DK055850 (NIH)
Record Dates: First submitted 2003-08-29; First posted 2003-09-01 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Growth Hormone; Diet Therapy

INTERVENTIONS:
Drug: recombinant human growth hormone
Behavioral: diet modification

SUMMARY:
This is a double-blind randomized controlled study on the clinical and metabolic effects and underlying gut mucosal mechanisms of modified diet, with or without recombinant human growth hormone, in adults with severe short bowel syndrome dependent upon parenteral nutrition. Clinical endpoints include ability to wean patients from parenteral feeding, metabolic endpoints include gut nutrient absorptive function and molecular endpoints include expression of growth factors and nutrient transporters in small bowel and colonic mucosa. The 6-month study is performed, in part, in the General Clinical Research Center for inpatient stays and outpatient visits.

DETAILED DESCRIPTION:
This is a double-blind randomized controlled study on the clinical and metabolic effects and underlying gut mucosal mechanisms of modified diet, with or without recombinant human growth hormone, in adults with severe short bowel syndrome dependent upon parenteral nutrition. Clinical endpoints include ability to wean patients from parenteral feeding, metabolic endpoints include gut nutrient absorptive function and molecular endpoints include expression of growth factors and nutrient transporters in small bowel and colonic mucosa. The 6-month study is performed, in part, in the General Clinical Research Center for inpatient stays and outpatient visits.

ELIGIBILITY:
* Parenteral nutrition-dependent adults with short gut syndrome.
* Patients must not have diabetes mellitus or active malignancy within the past 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 1996-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Ziegler, MD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States